CLINICAL TRIAL: NCT03624764
Title: A Randomized Comparative Study of Assisted Promontofixation Using Glue Versus Promontofixation Using Threads
Brief Title: Assisted Promontofixation Using Glue Versus Promontofixation Using Threads (PROCOL)
Acronym: PROCOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Beau Soleil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016- A01387-44
Record Dates: First submitted 2018-06-19; First posted 2018-08-10 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Prolapse
Keywords: promontofixation; prolapse surgery
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Promontofixation using glue (Experimental): Patients in this arm will have a laparoscopic promontofixation using a biocompatible cyanoacrylate adhesive replacing some sutures to maintain the strips.
  Interventions: Procedure: Laparostopic promontofixation using surgical glue
- Promontofixation using threads (Active Comparator): Patients in this arm will have a laparoscopic promontofixation using sutures with threads to maintain the strips.
  Interventions: Procedure: Laparostopic promontofixation using threads

INTERVENTIONS:
Procedure: Laparostopic promontofixation using surgical glue — The technique involves implanting a prosthetic tissue (tape) between the bladder and the vagina, suspending the cervix or the vagina affectionately, associated or not with a posterior strip placed between the rectum and the vagina fixed on the small pelvis muscles. Each strip is held by the surgical glue (cyanoacrylate biocompatible adhesive)
  Arms: Promontofixation using glue
Procedure: Laparostopic promontofixation using threads — The technique involves implanting a prosthetic tissue (tape) between the bladder and the vagina, suspending the cervix or the vagina affectionately, associated or not with a posterior strip placed between the rectum and the vagina fixed on the small pelvis muscles. Each strip is held by sutures with threads
  Arms: Promontofixation using threads

SUMMARY:
The treatment of gynecological prolapse (organ removal) can be done by laparoscopy or vaginally. Laparoscopy is used in 1 out of 2 cases, but learning is difficult and operation time is long. One of the technical difficulties is related to the sutures to the threads. Some surgeons therefore use a glue to fix prosthetic reinforcements more easily and quickly, but this sizing technique has only been evaluated very little. Our study proposes to compare the technique of suture with the thread at the gluing of the prostheses in order to validate the merits of this new technique

DETAILED DESCRIPTION:
Laparoscopic promontofixation is a surgical technique considered by some as the reference technique. Its difficulty of learning and the duration of operation are factors limiting its diffusion. The use of cyanoacrylate glue is proposed to simplify the procedure, without there being any comparative studies between the sutures over and the sizing of prosthetic reinforcements.

The main objective of the study is to compare the operative time of promontofixation by coelioscopy with suture using threads to promontofixation using glue.

Secondary objectives are the comparison between the two groups of complications per and postoperative, objective anatomical results and functional results of the tissue reaction judged by clinical examination (palpation) and ultrasound and direct cost.

ELIGIBILITY:
Inclusion Criteria:

1. Age> 40 years
2. Surgical indication of prolapse cure by promontofixation
3. Valid social insurance
4. French spoken and written
5. Informed consent signed
6. No exclusion criteria

Exclusion Criteria:

1. Concomitant rectopexy
2. Concomitant Hysterectomy
3. Associated surgical procedure not compatible with measurement of operative time
4. Refusal to participate in the study
5. Pregnant or lactating woman (Article L 1121-5 of the french code of public health)
6. Vulnerable persons (Article L 1121-6 of the french code of public health)
7. Majors subject to legal protection or unable to express their consent (Article 1121-8 of the CSP)
8. Participation in another protocol for less than 3 months
9. Patient does not have all the inclusion criteria.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-01-04 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2020-01-04 (Actual)

PRIMARY OUTCOMES:
Operative time | one day
  The time elapsed between incision and closure

SECONDARY OUTCOMES:
Collection of intra-operative complications | one day
  Collection of all the complications during the surgery (visceral wound, peroperative bleeding, other)
Collection of per-operative complications | one day
  Collection of the per-operative complications: pain at day 0 and day 1 (using the visual analog scale), urinary retention, postoperative haemorrhage or hematoma, fever> 38 ° 48 h after surgery, other complication
Collection of complications at 6 weeks | 6 weeks
  Pain by the Visuel Analog Scale, emergency consultation or generalist, rehospitalization / Reintervention, other complications
Tolerance of the prosthesis | 6 weeks
  Classification of the complications related to the insertion of protheses (from the International Urogynecological Association)
Tolerance of the prosthesis | 6 months
  Classification of the complications related to the insertion of protheses (from the International Urogynecological Association)
Tolerance of the prosthesis | 12 months
  Classification of the complications related to the insertion of protheses (from the International Urogynecological Association)
Objective anatomical results at 6 weeks | Before surgery
  International Continence Society - Pelvic organe Prolapse - Quantification (POP Q scale): stage 0 (no prolapse is demonstrated) to stage 4 (vaginal eversion is essentially complete)
Objective anatomical results at 6 months | 6 months after surgery
  International Continence Society - Pelvic organe Prolapse - Quantification (POP Q scale): stage 0 (no prolapse is demonstrated) to stage 4 (vaginal eversion is essentially complete)
Objective anatomical results at 12 month | 12 months after surgery
  International Continence Society - Pelvic organe Prolapse - Quantification (POP Q scale): stage 0 (no prolapse is demonstrated) to stage 4 (vaginal eversion is essentially complete)
Quality of life: pelvic floor distress | Before the surgery
  The Pelvic Floor Distress Inventory-20 questionnary: it is both a symptom inventory and a measure of the degree of bother and distress (quality-of-life) caused by pelvic floor symptoms.The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300. The 3 scales include questions taken from the following widely used outcome measures: Urinary Distress Inventory - 6 questions, Pelvic Organ Prolapse Distress Inventory - 6 questions, and Colorectal-Anal Distress Inventory - 8 questions
Quality of life: pelvic floor distress | 6 months after the surgery
  The Pelvic Floor Distress Inventory-20 questionnary. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300. The 3 scales include questions taken from the following widely used outcome measures: Urinary Distress Inventory - 6 questions, Pelvic Organ Prolapse Distress Inventory - 6 questions, and Colorectal-Anal Distress Inventory - 8 questions
Quality of life: pelvic floor distress | 12 months after the surgery
  The Pelvic Floor Distress Inventory-20 questionnary. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300. The 3 scales include questions taken from the following widely used outcome measures: Urinary Distress Inventory - 6 questions, Pelvic Organ Prolapse Distress Inventory - 6 questions, and Colorectal-Anal Distress Inventory - 8 questions

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Courtieu, Principal Investigator — Clinqieu Beau Soleil
Locations (1):
- Clinique Beau Soleil, Montpellier, France

IPD SHARING:
Plan to Share IPD: No